CLINICAL TRIAL: NCT00871156
Title: Safety, Tolerability, and Pharmacokinetic Study of Concomitant Chloroquine and Tafenoquine in Healthy Volunteers
Brief Title: Tafenoquine/Chloroquine DDI Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 106491
Record Dates: First submitted 2009-03-23; First posted 2009-03-30 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Malaria
Keywords: Drug-Drug Interaction
MeSH Terms: conditions — Malaria | interventions — Chloroquine; tafenoquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Active Comparator): Tafenoquine + Chloroquine vs. Chloroquine alone
  Interventions: Drug: Chloroquine, Tafenoquine
- Part 2 (Placebo Comparator): Chloroquine alone, Tafenoquine alone or Chloroquine+Tafenoquine
  Interventions: Drug: Chloroquine, Tafenoquine; Drug: Placebo

INTERVENTIONS:
Drug: Chloroquine, Tafenoquine — Chloroquine and Tafenoquine
  Other Names: Tafenoquine; Chloroquine
Drug: Placebo — Placebo
  Other Names: Placeob
  Arms: Part 2

SUMMARY:
DDI study of Tafenoquine and Chloroquine

DETAILED DESCRIPTION:
Safety, Tolerability, and Pharmacokinetic Study of Concomitant Chloroquine and Tafenoquine in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECGs. A subject with a clinical abnormality or laboratory parameters outside the reference range may be included only if the Investigator and GSK medical monitor agree that the abnormality will not introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential or of child-bearing potential if has a negative urine pregnancy test at screening and Day -1, and agrees to use agreed upon contraception methods until 56 days after stopping study drug.
* Body weight >=60 kg (132 pounds) and BMI within the range 19-32 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* A positive urine drug/alcohol screen at screening or Day -1.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of illicit drug abuse within 6 months prior to screening.
* History of regular alcohol consumption within 6 months of the study
* Subjects who are unwilling to comply with the lifestyle guidelines required.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of sensitivity to any of the study medications or their components.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Lactating females.
* Subject is mentally or legally incapacitated.
* A positive HIV antibody, Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject's systolic blood pressure is outside the range of 90-150mmHg or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects and 45-100bpm for male subjects at screening and Day -1.
* Cardiac conduction abnormalities as specified inprotocol
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* History of angina, ischemic heart disease, myocardial infarction, or clinically significant arrhythmia.
* History of epilepsy, convulsions or psychological disorders.
* History of porphyria.
* AST, ALT or alkaline phosphatase >1.5 times the upper limit of normal and/or total bilirubin level outside the normal range at screening. A single repeat is allowed for eligibility determination.
* Documented Glucose-6-phosphate dehydrogenase (G6PD) deficiency, determined by a quantitative assay of enzyme activity.
* History of hemoglobinopathy; or current or past history of methemoglobinemia or methemoglobin percentage above the reference range at screening.
* History of previous eye surgery involving the retina, Lasik surgery within 90 days, or retinal/corneal abnormalities.
* Any clinically significant abnormalities on the screening Humphrey 10-2 visual field test.
* Best corrected visual acuity worse than 0.3 logMAR (20/40 Snellen equivalent) (i.e., 20/40 or better vision will be allowed on study).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-03-24 (Actual); Primary Completion 2009-08-26 (Actual); Study Completion 2009-08-26 (Actual)

PRIMARY OUTCOMES:
TQ and Chloroquine (Day 2): AUC(0-tau), Cmax and Tmax | 56 days
CQ and TQ (Day 3): AUC(0-tau), AUC(0-inf), Cmax, Tmax and t1/2 | 56 days
AEs, vital signs, 12-lead ECGs, telemetry, clinical laboratory and ophthalmic assessments | 56 days

SECONDARY OUTCOMES:
QTcF, QT, QRS, RR and HR as assessed by 12-lead ECG | 56 Days
Changes from baseline in QTcF | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Background] Miller AK, Harrell E, Ye L, Baptiste-Brown S, Kleim JP, Ohrt C, Duparc S, Mohrle JJ, Webster A, Stinnett S, Hughes A, Griffith S, Beelen AP. Pharmacokinetic interactions and safety evaluations of coadministered tafenoquine and chloroquine in healthy subjects. Br J Clin Pharmacol. 2013 Dec;76(6):858-67. doi: 10.1111/bcp.12160. PMID 23701202
- See also: Results for study 106491 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/106491?search=study&study_ids=106491#rs